CLINICAL TRIAL: NCT06109493
Title: Effects of an ACT-based Psychological Treatment in Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Fundación Renal Iñigo Alvarez De Toledo (Other); Centro de Enseñanza Superior Cardenal Cisneros (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC040-23_FJD-FRIAT
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Diseases; Depression
MeSH Terms: conditions — Renal Insufficiency, Chronic; Depression

STUDY DESIGN:
Intervention Model Description: Randomization assigned participants to 2 arms:
  * ACT group
  * Waiting list
Who Masked: Participant
Masking Description: Participants did not know that two different treatments were delivered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT group (Experimental): 8 individual weekly sessions which included ACT methods
  Interventions: Behavioral: ACT
- Waiting list (No Intervention): Participants assigned to Waiting List arm waited for 5 months before receiving treatment

INTERVENTIONS:
Behavioral: ACT — Acceptance and Commitment Therapy methods were focused on promoting Values clarification, Acceptance, Cognitive defusion, Committed action and Flexible attention to the present moment, and included methods such as the Garden Metaphor, Funeral exercise or Mindfulness training.
  Arms: ACT group

SUMMARY:
Investigation of the efficacy of Acceptance and Commitment Therapy (ACT) for the psychological treatment of patients with chronic kidney disease.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

The clinical trial will include a control group (waiting list).

Patients who meet eligibility requirements will be assigned to control group or intervention group.

Psychological intervention will consist in an 8-session individual face-to-face delivered ACT-based treatment.

The participants will be assessed through self-report instruments before and after treatment and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease on haemodialysis
* Older than 18 years-old
* At least 3 months on haemodialysis
* HADS Global Scale Score ≥14

Exclusion Criteria:

* Diagnosis of severe or chronic mental disorder, mental retardation and cognitive impairment, or disabling illness.
* Antidepressant drugs consume
* Insufficient understanding of Spanish.
* Patients who are in the Advanced Chronic Kidney Disease Unit
* Receiving other psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in emotional distress assessed through Hospital Anxiety and Depression Scale (HADS) | Change from Baseline Emotional Distress at 5 months
  HADS assesses anxiety, depression and emotional distress. It is a 14-item four-point Likert-type scale. Scores range between 0 and 42. Higher the score in the overall score indicate higher levels of emotional distress and worse outcome.

SECONDARY OUTCOMES:
Change in Simplified Medication Adherence Questionnaire (SMAQ) | Change from Baseline Adherence at 5 months
  SMAQ assesses adherence to medication. It is a 6-item questionnaire that evaluates different aspects of patient compliance with treatment: forgetfulness, routine, adverse effects, and omissions. A patient is classified as non-compliant if he/she responds to any of the questions with a non-adherence answer, and in terms of quantification, if the patient has lost more than two doses during the last week or has not taken medication during more than two complete days during the last three months.
Change in COOP/WONCA questionnaire | Change from Baseline health related Quality of Life at 5 months
  COOP/WONCA assesses health related Quality of Life (HRQOL). It was selected the 7-item five-point Likert-type version of the scale. Scores range between 0 and 35. Higher scores indicate lower levels of HRQOL and worse outcome.
Change in Acceptance and Action Questionnaire in the context of Haemodialysis (CAAH-II) | Change from Baseline psychological inflexibility at 5 months
  Acceptance and Action Questionnaire' assesses psychological inflexibility. It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher scores indicate higher levels of psychological inflexibility and worse outcome.
Change in coping skills assessed through coping strategies inventory -short form (CSI-SF) | Change from Baseline coping strategies at 5 months
  CSI-SF is a 15-item, five-point Likert-type scale which includes four subscales: Problem Focused Engagement (PFE), Problem Focused Disengagement (PFD), Emotion Focused Engagement (EFE) and Emotion Focused Disengagement (EFD).
Change in mood assessed through Daylio App | Change from Baseline mood at 5 months
  Daylio is a mobile app which allows daily assessing mood through emoticons which will be transformed into a five-point Likert-type scale. Scores range between 1 and 5. Higher scores indicate higher better mood and better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, Ph.D., Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Fundación Renal Iñigo Alvarez de Toledo, Madrid, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06109493/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06109493/ICF_001.pdf